CLINICAL TRIAL: NCT05529862
Title: Trans-RosaLEE Study: a Biomarker-directed, Translational Study of High-throughput Molecular Profiling of HR+/HER2- Metastatic Breast Cancer Treated With Endocrine Therapy and Ribociclib.
Brief Title: Trans-RosaLEE Study: a Biomarker-directed, Translational Study
Acronym: TransRosaLEE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TransRosaLEE-IPC 2021-075
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Advanced or Metastatic Breast Cancer (BC)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally advanced or metastatic Breast Cancer Women (Experimental): Study Procedures:
  * Additional tumour sampling during the pre-treatment biopsy scheduled as per routine care,
  * A post-treatment tumour biopsy,
  * One pre-treatment and one post-treatment blood sampling.
  Interventions: Genetic: Pre-treatment biopsy; Genetic: Post treatment biopsy; Genetic: Pre treatment blood sampling; Genetic: Post treatment blood sampling

INTERVENTIONS:
Genetic: Pre-treatment biopsy — Pre-treatment fragments will be collected during the biopsy visit organised as part of routine medical practice, prior to the start of treatment with ribociclib + ET
Genetic: Post treatment biopsy — Post-treatment fragments will be collected during a biopsy visit specifically planned for Trans-RosaLEE study.
Genetic: Pre treatment blood sampling — Sampling of 4 EDTA Tubes (4ml) and 2 Streck tubes (10ml)
Genetic: Post treatment blood sampling — Sampling of 2 Streck tubes (10ml)

SUMMARY:
Hormone receptor (HR)-positive and HER2-negative (HR+/HER2-) metastatic/advanced breast cancer (mBC) is a major public health issue. During the last decades, a therapeutic challenge was to overcome the tumor's resistance to endocrine therapy (ET). Thanks to a better understanding of the molecular mechanisms of this resistance, effective new treatments have been developed, such as Kisqali® (ribociclib), a molecularly targeted therapy. This treatment blocks the growth and division of cancer cells by blocking proteins called CDK4/6 located inside the cell. This treatment, taken in combination with ET, blocks the harmful effect of hormones (estrogen) on cancer cell proliferation, and represent the standard first-line treatment of patients with HR+/HER2- mBC.

But, as with any treatment, it is expected that some patients will have a good response and their disease will be stabilized or even in remission, while other patients will not benefit from treatment and will relapse. In order to make progress, it is necessary to identify pre-therapeutic markers predictive of response to this treatment and the molecular mechanisms of this resistance set up by the tumor before or under the effect of the treatment.

The Trans-RosaLEE study aims to fill this gap by providing high-throughput molecular profiling (DNA and RNA) of a collection of tumor and blood samples from patients with RH+/HER2- mBC scheduled to start treatment with Kisqali® + ET. Samples will be collected just prior to initiation of therapy (pre-therapy) and just after discontinuation of therapy in the event of disease progression (post-therapy).

The main objectives of the TransRosaLEE study are :

* to determine if Kisqali® + ET treatment causes changes in the DNA and/or RNA genes of tumor;
* to identify whether there is a molecular signature that would predict clinical outcome of patients treated with Kisqali® + ET (tumor response, survival);
* to identify alterations in tumor's genes that could be targeted by a specific treatment and that would allow, in case of progression of the disease, to set up a new adapted treatment.

The TransRosaLEE study is a collaborative study between the Paoli-Calmettes Institute (France, Marseille) and the pharmaceutical group Novartis. It will take place in up to 90 healthcare institutions in France, and 241 patients will be enrolled. It is closely linked to the non-interventional study RosaLEE promoted by Novartis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in the RosaLEE study.
2. Patients having read and signed the ICF relative to Trans-RosaLEE.
3. Tumour material: primary and/or metastatic tumour sample, either available as frozen and collected within 3 months before V0, or newly collected before ribociclib + ET treatment initiation.

   Brain metastases and non-osteolytic bone metastases will be considered as non-collectable/biopsable.
4. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen.

Exclusion Criteria:

1. Not enrolled in RosaLEE.
2. Brain metastasis and non-osteolytic bone metastases as only metastatic sites, if no available frozen tumour sample already collected within 3 months before V0.
3. Tumour material not collected before ribociclib + ET initiation.
4. Person subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice), or unable to give their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Molecular alterations post- versus pre-treatment | At the date of first documented progression, assessed up to 54 months
  Occurrence of molecular alterations, including DNA copy number, gene mutations by WES and messenger RNA (mRNA) expression profiles by RNA-seq in paired post- versus pre-treatment samples.

SECONDARY OUTCOMES:
Molecular alterations associated with progression free survival | At 3 years after treatment initiation (Ribociclib+hormone therapy)
  Occurrence of molecular alterations in pre-treatment samples, such as DNA copy number alterations and mutational profiles analysed by WES, and mRNA expression profiles analysed by RNA-seq, associated with progression free survival.
Molecular alterations pre and post-treatment | At the date of first documented progression, assessed up to 54 months
  Occurrence of molecular alterations, including DNA copy number, gene mutations by WES and mRNA expression profiles by RNA-seq in the totality of pre- and post-treatment samples (paired and unpaired).
Pre treatment molecular alterations associated with tumor response | At 3 years after treatment initiation (Ribociclib+hormone therapy)
  Occurrence of molecular alterations in pre-treatment samples, such as DNA copy number alterations and mutational profiles analysed by WES and mRNA expression profiles analysed by RNA-seq, associated with tumour response according to RECIST 1.1 guidelines (complete and partial responses).
Molecular alterations therapeutically actionable | At the date of first documented progression, assessed up to 54 months
  Occurrence of molecular alterations in pre- and post-treatment samples, such as DNA copy number alterations and mutational profiles analysed by WES, which are therapeutically actionable according to the ESCAT scale.
Percentage of patients with molecular alterations therapeutically actionable | Through study completion, an average of 54 months
  Percentage of patients with molecular alterations such as DNA mutations and/or copy number alterations by WES, which are therapeutically actionable according to the ESCAT scale, in pre- and post-treatment samples.
Percentage of patients with modification of the therapeutic strategy derived from the molecular profiling | Through study completion, an average of 54 months
  Percentage of patients for which modification of the therapeutic strategy could have been derived from the molecular profiling of the post-treatment samples compared to that of the pre-treatment samples, according to the ESCAT scale.
IHC profile ER | At the date of first documented progression, assessed up to 54 months
  IHC profile ER of pre- and post-treatment samples.
IHC profile PgR | At the date of first documented progression, assessed up to 54 months
  IHC profile PgR of pre- and post-treatment samples.
IHC profile HER2 | At the date of first documented progression, assessed up to 54 months
  IHC profile HER2 of pre- and post-treatment samples.
Molecular subtypes PAM50 | At the date of first documented progression, assessed up to 54 months
  Molecular subtypes PAM50 of pre- and post-treatment samples.

CONTACTS AND LOCATIONS:
Overall Officials: François Bertucci, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No